CLINICAL TRIAL: NCT03013920
Title: A Prospective In-Vivo Human Pilot Study to Assess Confocal Laser Endomicroscopy Characteristics of Upper Tract Urothelial Carcinoma
Brief Title: CLE Characteristics of Upper Urinary Tract Urothelial Carcinoma
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof.dr. J.J.M.C.H. de la Rosette, Prof. dr. JJMCH de la Rosette, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2016_088
Record Dates: First submitted 2016-12-28; First posted 2017-01-09 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Urinary Tract Cancer; Urothelial Carcinoma; Ureter Cancer
Keywords: upper urinary tract cancer; confocal laser endomicroscopy; urothelial carcinoma
MeSH Terms: conditions — Urologic Neoplasms; Carcinoma, Transitional Cell; Ureteral Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — CLE images and histopathology
Oversight: Data Monitoring Committee: No

SUMMARY:
Rationale: Initial evaluation usually consists of cross sectional imaging of the urinary tract. When a suspect lesion is seen, an ureterorenoscopy is planned to visualize the lesion and to collect tissue for histopathology. These techniques are considered to be the gold standard in diagnosis of UTUC. CLE, a high resolution imaging technique that can be used in combination with endo-urological procedures, seems promising to improve diagnosis of urothelial cancer. CLE image characteristics for UTUC still have to be defined.

Objective: With this IDEAL stage 2b explorative pilot study the investigators aim to assess in-vivo CLE image characteristics of normal urothelium, benign urothelium and urothelial carcinoma (low-grade, high-grade or CIS) of the upper urinary tract by qualitatively comparing CLE images with both histopathology from diagnostic biopsies and pathology from the therapeutic radical nephroureterectomy. Secondary objectives are the development of an imaging atlas and to assess the technical feasibility and procedure related adverse events of CLE.

DETAILED DESCRIPTION:
This study is a prospective, mono-center observational human, in vivo pilot study to assess in-vivo CLE characteristics of normal urothelium, benign urothelium and urothelial carcinoma (low-grade, high-grade or CIS) of the upper urinary tract. Eligible patients have a suspect tumour in the upper urinary tract and are scheduled for a diagnostic URS. Eligible patients will be informed about this study by their urologist. Information about the study will be provided both verbally and in written form.

CLE images are recorded using a probe-based system (Cellvizio 100 series, Mauna Kea Technologies, Paris, France). The probe has a diameter of 0,85 mm, hereby enabling passage through the working channel of ureterorenoscope. It has a depth of tissue penetration of 50 µm, a field of view of 320 µm and a resolution of 3,5 µm. Images are collected at a scan rate of 12 frames per second. Using the Cellvizio Viewer system, we can observe mucosal microarchitecture with an increased field of view through mosaic post processing. This system also enables virtual staining of mucosal structures to further enhance tissue contrast.

A fluorescent contrast agent is needed to obtain CLE images. Fluorescein (fluoresceinedinatrium, Fresenius Kabi, Zeist, Nederland), a non-toxic and commonly used fluorescent dye will be administered through the working channel of the ureterorenoscope into the pyelocaliceal system (3 - 5 mL 0.1% fluorescein diluted in saline) and left indwelling for 5 minutes to stain the extracellular matrix.

In this study patients will undergo one CLE measurement during the planned diagnostic URS. We measure on average 2 regions of interest per patient. If a patient has multiple tumours we will do multiple measurements. The measurement duration per patient adds maximally 10 minutes during the URS. At a later stage two independent non-blinded observers will review the CLE images. The CLE images of the diagnostic URS are qualitatively compared with histopathology from diagnostic biopsies, and if performed also with pathology from the therapeutic nephroureterectomy.

Based on the UTUC diagnosis from the diagnostic URS, in general about one third of the patients are indicated for a therapeutic radical nephroureterectomy. The other two thirds of the UTUC patients are treated with endoscopic treatment. If patients undergo several ureterorenoscopies, they may be approached for CLE measurements at consecutive ureterorenoscopies.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years
* Suspect upper urinary tract urothelial carcinoma
* Scheduled for diagnostic URS
* Signed informed consent

Exclusion Criteria:

* Patients <18 years
* Patients with known allergy for fluorescein
* Possible pregnancy or lactating women
* Patients not eligible for radical treatment of UTUC
* No signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a suspect tumour in the upper urinary tract, who are planned for a diagnostic URS, are eligible for this study.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-08; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
In-vivo CLE measurements of normal urothelium and urothelial carcinoma (low-grade, high-grade or CIS) of the upper urinary tract | 3 years
  The CLE measurements are qualitatively correlated to the corresponding histopathology

CONTACTS AND LOCATIONS:
Overall Officials: Jean J de la Rosette, prof. dr., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liem EI, Freund JE, Baard J, de Bruin DM, Laguna Pes MP, Savci-Heijink CD, van Leeuwen TG, de Reijke TM, de la Rosette JJ. Confocal Laser Endomicroscopy for the Diagnosis of Urothelial Carcinoma in the Bladder and the Upper Urinary Tract: Protocols for Two Prospective Explorative Studies. JMIR Res Protoc. 2018 Feb 7;7(2):e34. doi: 10.2196/resprot.8862. PMID 29415874